CLINICAL TRIAL: NCT02605447
Title: A Prospective, Multicenter, Single-arm Study Designed to Assess the Safety of 3-month Dual Antiplatelet Therapy (DAPT) in Subjects at High Risk for Bleeding Undergoing Percutaneous Coronary Intervention (PCI) With the SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System
Brief Title: EVOLVE Short DAPT Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2073
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SYNERGY stent + 3 month DAPT (Experimental): Subject with implantation of at least one SYNERGY stent within the preceding 3 calendar days that takes the required dual antiplatelet therapy (3 months of P2Y12 inhibitor, 15 months of aspirin)
  Interventions: Drug: 3 months of dual antiplatelet therapy (DAPT); Device: SYNERGY Stent System

INTERVENTIONS:
Drug: 3 months of dual antiplatelet therapy (DAPT) — 3 months of P2Y12 inhibitor (clopidogrel, prasugrel or ticagrelor) plus 15-months of aspirin
Device: SYNERGY Stent System — SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System

SUMMARY:
The EVOLVE Short DAPT Study is a prospective, multicenter, single-arm study designed to assess the safety of 3-month DAPT in subjects at high risk for bleeding undergoing PCI with a SYNERGY Stent System.

DETAILED DESCRIPTION:
The primary objective of the EVOLVE Short DAPT Study is to assess the safety of 3-month dual antiplatelet therapy (DAPT) in subjects at high risk for bleeding undergoing percutaneous coronary intervention (PCI) with the SYNERGY Stent System.

The study will be conducted up to 120 sites worldwide in the United States, Europe, Japan, and Brazil with planned enrollment of up to 2,250 subjects. Clinical follow-up will be required at the following time points: 3 months, 6 months, 12 months and 15 months post index procedure.

Subjects must be treated with one of the following P2Y12 inhibitors (clopidogrel, prasugrel, or ticagrelor) for 3 months following the index procedure. Subjects must be treated with aspirin for the duration of the trial. The minimum daily maintenance dose of aspirin should be 75-100 mg.

Subjects are eligible for discontinuation of P2Y12 inhibitor at 3 months if they meet both of the following criteria: subject was treated with 3 months of study required antiplatelet therapy post index procedure; and subject was free from events (stroke, MI, PCI, coronary artery bypass graft [CABG], and stent thrombosis) between the index procedure and the 3 month visit.

Subjects are not eligible for discontinuation of P2Y12 inhibitor at 3 months if any of the following criteria are met: subject who experiences a stroke, MI, PCI, CABG and/or stent thrombosis, during the 0-3 month period (between the date of the index procedure and the date of the 3-month follow-up visit); or subject who is non-compliant with study required antiplatelet therapy during the 0-3 month period (between the date of the index procedure and the date of the 3-month follow-up visit); or subject judged inappropriate for discontinuation from P2Y12 inhibitor use at 3 months due to another condition requiring chronic P2Y12 inhibitor use.

All enrolled subjects who receive a SYNERGY stent must be followed at all milestones through 15-months, regardless of eligibility to discontinue P2Y12 inhibitor. Following the 3-month milestone, subjects who experience MI or stent thrombosis events should be treated per the investigator's discretion and should be followed through the 15-month visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is considered at high risk for bleeding, defined as meeting one or more of the following criteria at the time of enrollment:

   * ≥ 75 years of age and, in the opinion of the investigator, the risk of major bleeding associated with >3 months of DAPT outweighs the benefit,
   * need for chronic or lifelong anticoagulation,
   * history of major bleeding (severe/life threatening or moderate bleeding based on the GUSTO classification) within 12 months of the index procedure,
   * history of stroke (ischemic or hemorrhagic),
   * renal insufficiency (creatinine ≥2.0 mg/dl) or failure (dialysis dependent),
   * platelet count ≤100,000/μL
2. Subject must be at least 18 years of age
3. Subject must have had implantation of at least one SYNERGY stent within the preceding 3 calendar days
4. Subject must be able to take study required antiplatelet therapy (as required per protocol)
5. Subject is willing to comply with all protocol requirements, including agreement to stop taking P2Y12 inhibitor at the 3-month milestone, if eligible per protocol
6. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any study-specific procedures are performed
7. For subjects less than 20 years of age enrolled at a Japanese site, the subject/ the subject's legal representative must provide written informed consent before any study-specific tests or procedures are performed

Exclusion Criteria:

1. Subject with an indication for the index procedure of acute ST elevation MI (STEMI)
2. Subject with an indication for the index procedure of Non ST elevation MI (NSTEMI), based on the 3rd Universal MI definition
3. Subject with treatment with another coronary stent, other than SYNERGY, during the index procedure
4. Subject with planned staged procedures. (Note: Planned staged procedures are allowed if performed within 7 days and with only SYNERGY stents).
5. Subject has a known allergy to contrast (that cannot be adequately pre-medicated), the SYNERGY stent system or protocol-required concomitant medications (e.g., everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors and aspirin)
6. Subject with implantation of a drug-eluting stent within 9 months prior to index procedure
7. Subject previously treated at any time with intravascular brachytherapy
8. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
9. Subject is participating in an investigational drug or device clinical trial that has not reached its primary endpoint (Note: registry, observational, data collection studies are not exclusionary)
10. Subject intends to participate in an investigational drug or device clinical trial within 15 months following the index procedure (Note: registry, observational, data collection studies are not exclusionary)
11. Subject judged inappropriate for discontinuation from P2Y12 inhibitor use at 3 months, due to another condition requiring chronic P2Y12 inhibitor use
12. Subject with planned surgery or procedure necessitating discontinuation of P2Y12 inhibitor within 3 months following index procedure
13. Subject is a woman who is pregnant or nursing
14. Subject with a current medical condition with a life expectancy of less than 15 months
15. Target lesion(s) is located in the left main
16. Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate
17. Subject has unprotected left main coronary artery disease ( > 50% diameter stenosis)
18. Planned treatment of more than 3 lesion
19. Planned treatment of lesions in more than 2 major epicardial vessels
20. Target lesion(s) treated that involve complex bifurcation (i.e. bifurcation lesion requiring treatment with more than one stent)
21. Target lesion(s) is restenotic from a previous stent implantation
22. Target lesion(s) is located within a saphenous vein graft or an arterial graft
23. Target lesion(s) with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
24. Thrombus, or possible thrombus, present in the target vessel (by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2009 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, Principal Investigator — Columbia University Medical Center/ NewYork Presbyterian Hospital; Stephan Windecker, Prof, MD, Principal Investigator — INSELSPITAL - Universitätsspital Bern
Locations (110):
- United States (89):
  - Banner Good Samaritan Regional Medical Center, Phoenix, Arizona
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Baptist Health Medical Center (Little Rock), Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - USC Medical Center, Los Angeles, California
  - Cedars - Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - HCA Riverside Community Hospital, Riverside, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Foundation Hospital - San Francisco, San Francisco, California
  - John Muir Medical Center, Walnut Creek, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - Morton Plant Mease Healthcare System, Clearwater, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mediquest Research at Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Florida Hospital Heartland Medical Center, Sebring, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - University Hospital, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Edward Hospital, Naperville, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Franciscan St. Francis Hospital, Beech Grove, Indiana
  - Northern Indiana Research Alliance - Lutheran Hospital, Fort Wayne, Indiana
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - Jewish Hospital and St. Mary's Healthcare, Louisville, Kentucky
  - Cardiovascular Research, LLC, Shreveport, Louisiana
  - Maine Medical Center, Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - New York University Medical Center, New York, New York
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - University Medical Center-Greenville Memorial Hospital, Greenville, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - St. David's Round Rock Medical Center, Round Rock, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Aspirus Heart and Vascular Institute - Research and Education, Wausau, Wisconsin
- Brazil (2):
  - Instituto de Cardiologia Dante Pazzanese, São Paulo
  - Instituto do Coração (InCor), São Paulo
- Germany (4):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH, Bad Segeberg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Uni Jena, Jena
- Japan (10):
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - Kurume University Hospital, Kurume-shi
  - Osaka Saiseikai Nakatsu Hospital, Osaka
- P. Stradins University Hospital, Riga, Latvia
- Sweden (3):
  - Falu Lasarett, Falun
  - Karlstadt Central Hospital, Karlstad
  - Skane University Hospital, Malmo
- Hospital Cantonal Fribourg, Fribourg, Switzerland

REFERENCES:
- [Derived] Mihatov N, Kirtane AJ, Stoler R, Feldman R, Neumann FJ, Boutis L, Tahirkheli N, Kereiakes DJ, Toelg R, Othman I, Stein B, Allocco D, Windecker S, Yeh RW. Bleeding and Ischemic Risk Prediction in Patients With High Bleeding Risk (an EVOLVE Short DAPT Analysis). Am J Cardiol. 2023 Nov 15;207:370-379. doi: 10.1016/j.amjcard.2023.06.036. Epub 2023 Sep 29. PMID 37778226
- [Derived] Kirtane AJ, Stoler R, Feldman R, Neumann FJ, Boutis L, Tahirkheli N, Toelg R, Othman I, Stein B, Choi JW, Windecker S, Yeh RW, Dauerman HL, Price MJ, Underwood P, Allocco D, Meredith I, Kereiakes DJ. Primary Results of the EVOLVE Short DAPT Study: Evaluation of 3-Month Dual Antiplatelet Therapy in High Bleeding Risk Patients Treated With a Bioabsorbable Polymer-Coated Everolimus-Eluting Stent. Circ Cardiovasc Interv. 2021 Mar;14(3):e010144. doi: 10.1161/CIRCINTERVENTIONS.120.010144. Epub 2021 Mar 1. PMID 33641374
- [Derived] Balanescu DV, Aziz MK, Donisan T, Palaskas N, Lopez-Mattei J, Hassan S, Kim P, Song J, Ntim W, Cilingiroglu M, Marmagkiolis K, Iliescu C. Cancer treatment resumption in patients with new-generation drug-eluting stents. Coron Artery Dis. 2021 Jun 1;32(4):295-301. doi: 10.1097/MCA.0000000000000986. PMID 33196581
- [Derived] Mauri L, Kirtane AJ, Windecker S, Yeh RW, Dauerman HL, Price MJ, Christen T, Allocco DJ, Meredith IT, Kereiakes DJ. Rationale and design of the EVOLVE Short DAPT Study to assess 3-month dual antiplatelet therapy in subjects at high risk for bleeding undergoing percutaneous coronary intervention. Am Heart J. 2018 Nov;205:110-117. doi: 10.1016/j.ahj.2018.08.004. Epub 2018 Aug 17. PMID 30218844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2009 subjects enrolled at 110 centers in USA, Japan, Germany, Sweden, Brazil, Latvia and Switzerland between 16 February 2016 and 30 March 2018.
Pre-assignment Details: 2009 patients are enrolled, but 522 patients did not stop the DAPT therapy. Therefore 1487 patients are counted as eligible for the study endpoints.
Groups:
- SYNERGY Stent + 3 Month DAPT: Subject with implantation of at least one SYNERGY stent within the preceding 3 calendar days that takes the required dual antiplatelet therapy (3 months of P2Y12 inhibitor, 15 months of aspirin)
  3 months of dual antiplatelet therapy (DAPT): 3 months of P2Y12 inhibitor (clopidogrel, prasugrel or ticagrelor) plus 15-months of aspirin
  SYNERGY Stent System: SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System
  2009 patients are enrolled, but 522 patients did not stop the DAPT therapy. Therefore 1487 patients are counted as eligible for the study endpoints.
Period: Overall Study
Arm/Group | SYNERGY Stent + 3 Month DAPT
Started | 1487
Completed | 1385
Not Completed | 102
Not completed — Death | 66
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 24
Not completed — Withdrawal by Subject | 10
Not completed — Not disclosed | 1

BASELINE CHARACTERISTICS:
Population: 2009 patients are enrolled, but 522 patients did not stop the DAPT therapy. Therefore 1487 patients are counted as eligible for the study endpoints.
Arm/Group | SYNERGY Stent + 3 Month DAPT
Number analyzed (Participants) | 1487
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 506
  Male | 981
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 7
  Asian | 130
  Black, African Heritage | 70
  Caucasian | 1159
  Hispanic or Latino | 45
  Native Hawaian or other Pacific Islander | 1
  Other | 14
  Not Disclosed | 66
Region of Enrollment [Number; unit: participants]
  Latvia | 25
  Sweden | 21
  United States | 1177
  Japan | 117
  Brazil | 29
  Switzerland | 13
  Germany | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Death or Myocardial Infarction (MI)
Description: Rate of death or myocardial infarction
Time Frame: 3 to 15 months
Population: 2009 patients are enrolled, but 522 patients did not stop the DAPT therapy. Therefore 1487 patients are counted as eligible for the study endpoints. Among these, 30 patients who didn't have sufficient follow-up nor an event were not eligible for analysis of the CEC confirmed major adverse events from 3-month visit to 365 days post 3-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | SYNERGY Stent + 3 Month DAPT
Number analyzed (Participants) | 1457
Participants | 84

2. Primary Outcome: Number of Participants Who Experienced Stent Thrombosis (ST)
Description: Rate of stent thrombosis: definite + probable, using the Academic Research Consortium (ARC) definition Confirmed/Definite (is considered either angiographic confirmed or pathologic confirmed) Probable
  Clinical definition of probable stent thrombosis is considered to have occurred in the following cases:
  * Any unexplained death within the first 30 days
  * Irrespective of the time after the index procedure and MI in the absence of any obvious cause which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis Possible Clinical definition of possible stent thrombosis is considered to have occurred with any unexplained death beyond 30 days.
Time Frame: 3 to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYNERGY Stent + 3 Month DAPT
Number analyzed (Participants) | 1457
Participants | 3

3. Secondary Outcome: Number of Participants Who Experienced Major Bleeding
Description: Rate of Bleeding, per Bleeding Academic Consortium definition (BARC2, 3a, 3b, 3c, 4, 5a and 5b)
  * Type 0: No Bleeding
  * Type 1: Bleeding that is not actionable and does not cause the patient to seek treatment
  * Type 2: Any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional
  * Type 3a: Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
  * Type 3b: Overt bleeding plus hemoglobin drop ≥5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
  * Type 3c: Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision
  * Type 4: CABG-related bleeding within 48 hours
  * Type 5a: Probable fatal bleeding
  * Type 5b: Definite fatal bleeding
Time Frame: 3 to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SYNERGY Stent + 3 Month DAPT
Number analyzed (Participants) | 1457
Participants | 103

ADVERSE EVENTS:
Time Frame: Study start to end of study (15 month)
Description: 2009 patients are enrolled, but 522 patients did not stop the DAPT therapy. Therefore 1487 patients are counted as eligible for the study endpoints.
  66 patients passed away between 3 month and end of study. Patients who passed away before 3 month are not considered eligible for the primary endpoint analysis. Death for unknown reason are reported as Death or cardiac Death
Arm/Group | SYNERGY Stent + 3 Month DAPT
All-Cause Mortality (participants affected / at risk) | 66/1487
Serious Adverse Events (participants affected / at risk) | 607/1487
Other Adverse Events (participants affected / at risk) | 100/1487
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGY Stent + 3 Month DAPT (N=1487)
Anaemia (Blood and lymphatic system disorders) | 20 (22)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 8 (9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Total (Blood and lymphatic system disorders) | 38 (43)
Acute coronary syndrome (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 21 (24)
Acute right ventricular failure (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 33 (36)
Angina unstable (Cardiac disorders) | 17 (17)
Aortic valve disease (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 16 (17)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 60 (73)
Atrial flutter (Cardiac disorders) | 5 (5)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 5 (5)
Bradycardia (Cardiac disorders) | 8 (8)
Cardiac arrest (Cardiac disorders) | 9 (9)
Cardiac failure (Cardiac disorders) | 15 (15)
Cardiac failure acute (Cardiac disorders) | 6 (6)
Cardiac failure chronic (Cardiac disorders) | 10 (15)
Cardiac failure congestive (Cardiac disorders) | 47 (61)
Cardiac perforation (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 3 (3)
Cardiomyopathy (Cardiac disorders) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 2 (2)
Cardiorenal syndrome (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 18 (20)
Coronary artery dissection (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 10 (10)
Extrasystoles (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 4 (5)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 3 (3)
Sinus arrest (Cardiac disorders) | 3 (3)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3)
Total (Cardiac disorders) | 264 (378)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1)
Total (Congenital, familial and genetic disorders) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
Total (Ear and labyrinth disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Steroid withdrawal syndrome (Endocrine disorders) | 1 (1)
Total (Endocrine disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Total (Eye disorders) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Enteritis (Gastrointestinal disorders) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Faecaloma (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 20 (21)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 3 (3)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (3)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Total (Gastrointestinal disorders) | 88 (104)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Cardiac death (General disorders) | 1 (1) — Sites are instructed to report the adverse event leading to death, however in some instances sites could only report death due to unknown reason.
Catheter site haematoma (General disorders) | 7 (7)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 13 (13)
Coronary artery restenosis (General disorders) | 1 (1)
Death (General disorders) | 6 (6) — Sites are instructed to report the adverse event leading to death, however in some instances sites could only report death due to unknown reason.
Device lead damage (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 41 (47)
Peripheral swelling (General disorders) | 2 (3)
Pyrexia (General disorders) | 4 (4)
Strangulated hernia (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 1 (1)
Total (General disorders) | 85 (96)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Total (Hepatobiliary disorders) | 13 (17)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Kidney transplant rejection (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Total (Immune system disorders) | 6 (6)
Abdominal abscess (Infections and infestations) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 5 (5)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (2)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Diabetic gangrene (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3)
Endocarditis (Infections and infestations) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4)
Herpes zoster (Infections and infestations) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 10 (10)
Intervertebral discitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 2 (2)
Perirectal abscess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (2)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 34 (38)
Postoperative wound infection (Infections and infestations) | 1 (1)
Proteus infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 19 (22)
Septic shock (Infections and infestations) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Total (Infections and infestations) | 107 (147)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 14 (17)
Urosepsis (Infections and infestations) | 4 (4)
Viral infection (Infections and infestations) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Total (Injury, poisoning and procedural complications) | 72 (84)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 10 (11)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 12 (12)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3)
Blood pressure decreased (Investigations) | 1 (1)
Computerised tomogram abdomen abnormal (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Total (Investigations) | 6 (6)
Troponin increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 3 (3)
Gout (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Total (Metabolism and nutrition disorders) | 18 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hungry bone syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Total (Musculoskeletal and connective tissue disorders) | 33 (38)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Total (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 (54)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 8 (9)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 13 (14)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Dementia (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2)
Dementia with Lewy bodies (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Dysarthria (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 5 (5)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 2 (2)
Migraine (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Myasthenic syndrome (Nervous system disorders) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 6 (6)
Sciatica (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 10 (11)
Tension headache (Nervous system disorders) | 1 (1)
Total (Nervous system disorders) | 80 (95)
Transient ischaemic attack (Nervous system disorders) | 7 (7)
Mental status changes (Psychiatric disorders) | 3 (3)
Neurosis (Psychiatric disorders) | 1 (1)
Total (Psychiatric disorders) | 4 (4)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Diabetic end stage renal disease (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (9)
Nephrolithiasis (Renal and urinary disorders) | 6 (6)
Obstructive uropathy (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (5)
Renal failure acute (Renal and urinary disorders) | 35 (39)
Renal failure chronic (Renal and urinary disorders) | 11 (11)
Renal haemorrhage (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Total (Renal and urinary disorders) | 70 (84)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (6)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Total (Reproductive system and breast disorders) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (18)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Total (Respiratory, thoracic and mediastinal disorders) | 73 (86)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Total (Skin and subcutaneous tissue disorders) | 3 (3)
Aortic aneurysm (Vascular disorders) | 5 (5)
Aortic dissection (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 5 (5)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Femoral artery aneurysm (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Hypertensive crisis (Vascular disorders) | 6 (8)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 10 (11)
Intermittent claudication (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 5 (6)
Peripheral artery stenosis (Vascular disorders) | 3 (4)
Peripheral ischaemia (Vascular disorders) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 4 (4)
Shock (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Total (Vascular disorders) | 54 (68)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGY Stent + 3 Month DAPT (N=1487)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Total (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Total (Cardiac disorders) | 3 (3)
Eye haemorrhage (Eye disorders) | 1 (1)
Total (Eye disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 4 (5)
Haematochezia (Gastrointestinal disorders) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 9 (9)
Total (Gastrointestinal disorders) | 22 (25)
Catheter site haematoma (General disorders) | 7 (7)
Catheter site haemorrhage (General disorders) | 3 (3)
Implant site haematoma (General disorders) | 1 (1)
Total (General disorders) | 11 (11)
Total (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 5 (6)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 3 (3)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Total (Injury, poisoning and procedural complications) | 23 (26)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Occult blood (Investigations) | 1 (1)
Total (Investigations) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Total (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Total (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 15 (18)
Total (Renal and urinary disorders) | 15 (18)
Total (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 (28)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Total (Respiratory, thoracic and mediastinal disorders) | 27 (30)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3 (3)
Total (Skin and subcutaneous tissue disorders) | 4 (4)
Bleeding varicose vein (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (3)
Haemorrhage (Vascular disorders) | 1 (1)
Total (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT02605447/Prot_SAP_000.pdf